CLINICAL TRIAL: NCT00258453
Title: Prospective, Multi-Center Survey Study of Children and Adolescents With Craniopharyngioma
Brief Title: Observation of Young Patients Who Are Undergoing Surgery for Craniopharyngioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: GPOH-CRANIOPHARYNGIOMA-2000; CDR0000450768 (Registry Identifier: PDQ (Physician Data Query)); EU-20537
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2007-10

CONDITIONS: Brain and Central Nervous System Tumors; Long-term Effects Secondary to Cancer Therapy in Children; Perioperative/Postoperative Complications; Psychosocial Effects of Cancer and Its Treatment; Weight Changes
Keywords: psychosocial effects of cancer and its treatment; long-term effects secondary to cancer therapy in children; perioperative/postoperative complications; weight changes; childhood craniopharyngioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Postoperative Complications; Body Weight Changes | interventions — Biopsy; Magnetic Resonance Spectroscopy; Psychiatric Rehabilitation; Radiotherapy

INTERVENTIONS:
Other: metabolic assessment
Other: physiologic testing
Procedure: biopsy
Procedure: computed tomography
Procedure: conventional surgery
Procedure: magnetic resonance imaging
Procedure: management of therapy complications
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Collecting information on how craniopharyngioma is diagnosed and treated may help doctors predict a patient's response to treatment and help plan the best treatment. It may also help identify the intermediate- and long-term effects of treatment.

PURPOSE: This clinical trial is collecting information on diagnosis, treatment, and quality of life of young patients who are undergoing surgery for craniopharyngioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify all applied therapy strategies in pediatric patients with craniopharyngioma.
* Correlate relapse status with different therapy strategies/modality in these patients.
* Determine the health status (i.e., ophthalmologic, neuropediatric, and endocrine findings) and the health-related quality of life of these patients after treatment.

Secondary

* Determine the incidence of craniopharyngioma in pediatric patients.
* Identify quality control measures for diagnosis and therapy in these patients.
* Improve long-term care through a standardized follow-up program in these patients.
* Determine the efficacy of endocrine substitution for postoperative hypopituitarism in these patients.
* Identify risk factors for developing obesity and correlate the neurotransmitter concentration of leptin and neuropeptide Y in cerebral spinal fluid, serum, and craniopharyngioma cystic fluid with the likelihood of developing obesity in these patients.
* Determine the incidence and extent of eating disorders in these patients.

OUTLINE: This is a multicenter study.

Patients undergo neurologic, endocrine, and ophthalmologic tests and anthropometric diagnostic measurements. Patients then undergo 1 of the following surgical procedures: total resection; incomplete, subtotal, or partial resection; biopsy; or cyst pressure release. Patients whose tumor relapses may undergo a second resection and/or radiotherapy.

Quality of life is assessed at baseline and then periodically thereafter.

After surgery, patients are followed periodically.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary craniopharyngioma by MRI and CT scan (initial diagnosis)

  * Patients with only cystic sellar or parasellar malformation (e.g., Rathke pouch cysts or suprasellar cysts) are allowed but will undergo observation only

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY: Not specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2001-05; Primary Completion 2007-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Mueller, MD, Study Chair — Klinikum Oldenburg
Locations (109):
- Austria (13):
  - Krankenhaus Dornbirn, Dornbirn
  - Landeskrankenhaus Feldkirch, Feldkirch-Tisis
  - Universitaet Kinderklinik, Graz
  - Innsbruck Universitaetsklinik, Innsbruck
  - Landeskrankenhaus Klagenfurt, Klagenfurt
  - LKH Leoben, Leoben
  - A. oe. Krankenhaus der Barmherzigen Schwestern Kinderabteilung, Linz
  - Landes-Kinderkrankenhaus, Linz
  - St. Johanns-Spital, Salzburg
  - Kardinal Schwarzenbersches Krankenhaus Betriebsgesellschraft mbH Kinderspital, Schwarzach
  - A. oe. Landeskrankenhaus Abt. fuer Kinderkrankheiten, Steyr
  - Allg. Krankenhaus der Stadt Wien Universitaets-Kinderklinik, Vienna
  - St. Anna Children's Hospital, Vienna
- Germany (88):
  - Kinderklinik - Universitaetsklinikum Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Caritas-Krankenhaus Bad Mergentheim, Bad Mergentheim
  - Klinikum am Bamberg, Bamberg
  - Klinikum Bayreuth, Bayreuth
  - Helios Klinikum Berlin, Berlin
  - Charite - Campus Charite Mitte, Berlin
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Evangelisches Krankenhauus Bielfeld, Biefeld
  - Kinderklinik der Universitaet Bonn, Bonn
  - Klinikum Bremen-Mitte, Bremen
  - Allgemeinen Krankenhaus Celle Kinderklinik, Celle
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Klinikum Coburg, Coburg
  - Kliniken der Stadt Koeln gGmbH - Kinderkrankenhaus Riehl, Cologne
  - Children's Hospital, Cologne
  - Carl - Thiem - Klinkum Cottbus, Cottbus
  - Vestische Kinderklinik Universitaetsklinik Witten/Herdecke, Datteln
  - Klinikum Lippe - Detmold, Detmold
  - Staedtisches Krankenhaus Dresden - Neustadt, Dresden
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Klinikum Duisburg, Duisburg
  - Klinikum Erfurt, Erfurt
  - Universitaets - Kinderklinik, Erlangen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitaetskinderklinik - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Kinderklinik, Giessen
  - Universitaetsklinikum Goettingen, Göttingen
  - Universitats - Kinderklinik, Greiswald
  - Kreiskrankenhaus Gummersbach GMBH, Gummersbach
  - Universitaetsklinikum Halle, Halle
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Kreskrankenhaus Kinderabteilung, Heide
  - Universitaets-Kinderklinik Heidelberg, Heidelberg
  - SLK - Kliniken Heilbronn GmbH - Klinikum am Gesundbrunnen, Heilbronn
  - Gemeinschaftskrankenhaus, Herdecke
  - Staedtisches Krankenhaus Hildesheim, Hildesheim
  - Universitaetsklinikum des Saarlandes, Homburg
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Universitaets - Kinderklinik, Jena
  - Municipal Hospital Complex of the University, Kaiserslautern
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Klinikum Kassel, Kassel
  - Staedtisches Krankenhaus Kiel, Kiel
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Klinikum Kemperhof Koblenz, Koblenz
  - Klinik Konstanz, Konstanz
  - Klinikum Krefeld GmbH, Krefeld
  - Kinderkrankenhaus St. Marien, Landshut
  - Universitaets - Kinderklinik, Leipzig
  - St. Annastift Krankenhaus, Ludwigshafen
  - Universitaets - Kinderklinik - Luebeck, Lübeck
  - Universitatsklinikum der MA, Magdeburg
  - Johannes Gutenberg University, Mainz
  - Staedtisches Klinik - Kinderklinik, Mannheim
  - Universitaets - Kinderklinik, Marburg
  - Klinikum Minden, Minden
  - Krankenhaus Neuwerk Klinik fuer Kinder und Jugendmedizin, Mönchengladbach
  - Krankenhaus Muenchen Schwabing, Munich
  - Dr. von Haunersches Kinderspital der Universitaet Muenchen, Munich
  - Staedtisches Krankenhaus Muenchen - Harlaching, Munich
  - Klinik und Poliklinik fuer Kinder und Jugendmedizin - Universitaetsklinikum Muenster, Münster
  - Klinikum Neubrandenburg, Neubrandenburg
  - Lukaskrankenhaus Neuss, Neuss
  - Marienhaus Klinikum St. Elisabeth Neuwied, Neuwied
  - Cnopf'sche Kinderklinik, Nuremberg
  - Klinikum Nuernberg - Klinikum Sued, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - Marien Hospital, Osnabrück
  - Paracelsus - Klinik Osnabrueck, Osnabrück
  - Klinik St. Hedwig-Kinderklinik, Regensburg
  - Kinderklinik - Universitaetsklinikum Rostock, Rostock
  - Saarbrucker Winterbergkliniken, Saarbrücken
  - Johanniter-Kinderklinik, Sankt Augustin
  - Klinikum Schwerin, Schwerin
  - Kinderklink Siegen Deutsches Rotes Kreuz, Siegen
  - Olgahospital, Stuttgart
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Universitaetsklinikum Tuebingen, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - St. Marienhospital - Vechta, Vechta
  - Staedtisches Klinikum - Howedestrase, Vechta
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Reinhard-Nieter-Krankenhaus, Wilhelmshaven
  - Klinikum der Stadt Wolfsburg, Wolfsburg
  - Helios Kliniken Wuppertal University Hospital, Wuppertal
  - Universitaets - Kinderklinik Wuerzburg, Würzburg
- Lanssjukhuset Ryhov, Jönköping, Sweden
- Switzerland (7):
  - Kantonspital Aarau, Aarau
  - Universitaets-Kinderspital beider Basel, Basel
  - Ospedale "la Carita", Locarno, Locarno
  - Kinderspital Luzern, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - University Children's Hospital, Zurich

REFERENCES:
- [Result] Roth CL, Gebhardt U, Muller HL. Appetite-regulating hormone changes in patients with craniopharyngioma. Obesity (Silver Spring). 2011 Jan;19(1):36-42. doi: 10.1038/oby.2010.80. Epub 2010 Apr 8. PMID 20379145
- [Result] Muller HL, Gebhardt U, Schroder S, Pohl F, Kortmann RD, Faldum A, Zwiener I, Warmuth-Metz M, Pietsch T, Calaminus G, Kolb R, Wiegand C, Sorensen N; study committee of KRANIOPHARYNGEOM 2000/2007. Analyses of treatment variables for patients with childhood craniopharyngioma--results of the multicenter prospective trial KRANIOPHARYNGEOM 2000 after three years of follow-up. Horm Res Paediatr. 2010;73(3):175-80. doi: 10.1159/000284358. Epub 2010 Mar 3. PMID 20197669
- [Derived] Sowithayasakul P, Beckhaus J, Ozyurt J, Bison B, Friedrich C, Muller HL. Prolactin serum concentrations in childhood-onset craniopharyngioma patients. J Endocrinol Invest. 2025 Sep;48(9):2041-2051. doi: 10.1007/s40618-025-02622-4. Epub 2025 Jun 7. PMID 40481916
- [Derived] Mann-Markutzyk LV, Beckhaus J, Ozyurt J, Mehren A, Friedrich C, Muller HL. Daytime sleepiness and health-related quality of life in patients with childhood-onset craniopharyngioma. Sci Rep. 2025 Mar 19;15(1):9407. doi: 10.1038/s41598-025-94384-5. PMID 40108339
- [Derived] Wagener K, Beckhaus J, Boekhoff S, Friedrich C, Muller HL. Sporadic and neurofibromatosis type 2-associated meningioma in children and adolescents. J Neurooncol. 2023 Jul;163(3):555-563. doi: 10.1007/s11060-023-04344-0. Epub 2023 Jul 4. PMID 37402092
- [Derived] Beckhaus J, Friedrich C, Boekhoff S, Calaminus G, Bison B, Eveslage M, Timmermann B, Flitsch J, Muller HL. Outcome after pediatric craniopharyngioma: the role of age at diagnosis and hypothalamic damage. Eur J Endocrinol. 2023 Mar 2;188(3):lvad027. doi: 10.1093/ejendo/lvad027. PMID 36857103
- [Derived] Mehren A, Ozyurt J, Zu Klampen P, Boekhoff S, Thiel CM, Muller HL. Self- and informant-rated apathy in patients with childhood-onset craniopharyngioma. J Neurooncol. 2018 Oct;140(1):27-35. doi: 10.1007/s11060-018-2936-z. Epub 2018 Jul 3. PMID 29971569
- [Derived] Ozyurt J, Muller HL, Warmuth-Metz M, Thiel CM. Hypothalamic tumors impact gray and white matter volumes in fronto-limbic brain areas. Cortex. 2017 Apr;89:98-110. doi: 10.1016/j.cortex.2017.01.017. Epub 2017 Feb 3. PMID 28259055
- [Derived] Daubenbuchel AM, Hoffmann A, Eveslage M, Ozyurt J, Lohle K, Reichel J, Thiel CM, Martens H, Geenen V, Muller HL. Oxytocin in survivors of childhood-onset craniopharyngioma. Endocrine. 2016 Nov;54(2):524-531. doi: 10.1007/s12020-016-1084-5. Epub 2016 Sep 1. PMID 27585663
- [Derived] Hoffmann A, Warmuth-Metz M, Lohle K, Reichel J, Daubenbuchel AM, Sterkenburg AS, Muller HL. Fusiform dilatation of the internal carotid artery in childhood-onset craniopharyngioma: multicenter study on incidence and long-term outcome. Pituitary. 2016 Aug;19(4):422-8. doi: 10.1007/s11102-016-0722-5. PMID 27125511
- [Derived] Ozyurt J, Thiel CM, Lorenzen A, Gebhardt U, Calaminus G, Warmuth-Metz M, Muller HL. Neuropsychological outcome in patients with childhood craniopharyngioma and hypothalamic involvement. J Pediatr. 2014 Apr;164(4):876-881.e4. doi: 10.1016/j.jpeds.2013.12.010. Epub 2014 Feb 6. PMID 24507865
- [Derived] Roth CL, Enriori PJ, Gebhardt U, Hinney A, Muller HL, Hebebrand J, Reinehr T, Cowley MA. Changes of peripheral alpha-melanocyte-stimulating hormone in childhood obesity. Metabolism. 2010 Feb;59(2):186-94. doi: 10.1016/j.metabol.2009.06.031. Epub 2009 Sep 18. PMID 19766264